CLINICAL TRIAL: NCT00035321
Title: The Study of Olanzapine Plus Fluoxetine in Combination for Treatment-Resistant Depression Without Psychotic Features
Brief Title: The Study of Olanzapine Plus Fluoxetine in Combination for Treatment of Treatment Resistant Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6272; H6P-MC-HDAO
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2006-07-24 (Estimated); Status verified 2006-07

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Olanzapine; Fluoxetine

INTERVENTIONS:
Drug: Olanzapine
Drug: Fluoxetine

SUMMARY:
The purposes of this study are to determine:

* Whether olanzapine plus fluoxetine in combination will help patients with treatment-resistant major depression.
* The safety of olanzapine plus fluoxetine in combination, plus and any side effects that might be associated with the combination.
* The effectiveness of olanzapine plus fluoxetine compared to olanzapine and fluoxetine alone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 18 - 65 years of age.
* Each patient must have a level of understanding sufficient to perform all tests and examinations required by the protocol, and must be considered reliable according to the investigator's clinical judgement
* Patients must fulfill the criteria for recurrent MDD without psychotic features as defined by the DSM-IV, based on clinical assessment and confirmed by Structured Clinical Interview for DSM-IV Axis I Disorders - Clinical Version (SCID-I) plus the Major Depressive Disorder Specifiers included in the Research Version of the SCID-I. This includes at least one of the following diagnoses: 296.31, 296.32, and 296.33
* Female patients of childbearing potential must be using a medically accepted means of contraception throughout the course of the study. Use of any oral or injectable contraception must be initiated prior to visit 2
* Failure to achieve satisfactory antidepressant response to an adequate trial of an antidepressant (except fluoxetine), for at least 6 weeks at an acceptable dose or greater, occurring within the current episode of MDD

Exclusion Criteria:

* Treatment with a drug within the last 30 days that has not received regulatory approval at the time of study entry
* Exposure to OFC in a Lilly-sponsored clinical trial investigating OFC, and any patients historically failing to respond to olanzapine and fluoxetine in combination under any circumstance
* Persons who have previously entered any Lilly-sponsored study which was investigating olanzapine
* Female patients who are either pregnant or nursing
* Serious, unstable illnesses for which death is anticipated within 1 year of intensive care unit hospitalization for the disease is anticipated within 6 months. This includes hepatic (specifically any degree of jaundice), renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic diseases (specifically current agranulocytosis with an absolute neutrophil count < 500 mm_3)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2002-04; Study Completion 2005-07

PRIMARY OUTCOMES:
To assess the efficacy of up to 8 weeks of treatment with OFC versus olanzapine and fluoxetine monotherapies, in patients with recurrent MDD without psychotic features
who meet study criteria for TRD, as measured by last observation carried forward (LOCF) mean change from baseline to endpoint in the MADRS total score
Treatment-resistant depression will be defined as:historic failure to achieve satisfactory response to an antidepressant (other than fluoxetine) during the current MDD episode
when treated with an acceptable antidepressant drug and dose for at least 6 weeks
prospective failure to achieve a satisfactory response to fluoxetine monotherapy during the 8 week study lead-in phase

SECONDARY OUTCOMES:
To compare the efficacy, safety, and quality of life results of up to 8 weeks of OFC therapy(treatment phase) with fluoxetine and olanzapine monotherapies using the following assessments:
Onset of action as measured by time to achieve and initial response (greater than or equal to 25% reduction from baseline in MADRS total score
Efficacy in the treatment of co-morbid anxiety symptoms as measured by LOCF mean change from baseline to endpoint in Hamilton Psychiatric Rating Scale for Anxiety (HAM-A)total score
Study-defined response and remission rates including time to achieve a full response (defined as greater than or equal to 50% reduction in MADRS total score)
and time to achieve remission (defined as MADRS total score less than or equal to 10 at endpoint)
LOCF mean change from baseline to endpoint in Clinical Global Impression - Severity of Depression score
(CGI-Severity of Depression), individual MADRS questions,and HAM-A item scores
Repeated measures analyses of post-baseline MADRS and HAM-A total scores
The incidence and severity of treatment-emergent adverse events and EPS. The Barnes Akathisia Scale,Simpson-Angus Scale, and the Abnormal Involuntary Movement Scale (AIMS) will be used to assess EPS
The Brief Psychiatric Rating Scale (BPRS) to evaluate the emergence of psychosis
Changes in vital signs and weight, laboratory analytes, and electrocardiograms (ECG)),Quality of life as measured by the LOCF mean change from baseline to endpoint on the Sheehan Disability Scale (SDS) score and the Short Form 36 Health Survey
Additional secondary objectives are to assess the efficacy, safety, and quality of life results of up to 8 additional weeks of open-label OFC therapy (after the treatment phase)using the following measures:
LOCF mean change from baseline to endpoint in MADRS, HAM-A, and CGI-Severity of Depression scores and study-defined rates of response and remission
Safety as measured by the incidence and severity of treatment-emergent adverse events, and EPS using the Barnes Akithisia Scale, Simpson Angus Scale and the AIM
The BPRS to examine the emergence of psychosis
Changes in vital signs and weight, laboratory analytes, and ECG

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (33):
- United States (30):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oceanside, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Marcos, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torrance, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New London, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coral Springs, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., North Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St. Petersburg, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marietta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Libertyville, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oak Brook, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Orleans, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glen Burnie, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Westminster, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsfield, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clementon, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moorestown, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toms River, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dayton, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Medford, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salem, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sellersville, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lincoln, Rhode Island
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waukesha, Wisconsin
- Canada (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St. John's, Newfoundland and Labrador
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kingston, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St. John's

REFERENCES:
- [Derived] Houston JP, Kohler J, Bishop JR, Ellingrod VL, Ostbye KM, Zhao F, Conley RR, Poole Hoffmann V, Fijal BA. Pharmacogenomic associations with weight gain in olanzapine treatment of patients without schizophrenia. J Clin Psychiatry. 2012 Aug;73(8):1077-86. doi: 10.4088/JCP.11m06916. PMID 22967772
- [Derived] Houston JP, Lau K, Aris V, Liu W, Fijal BA, Heinloth AN, Perlis RH. Association of common variations in the norepinephrine transporter gene with response to olanzapine-fluoxetine combination versus continued-fluoxetine treatment in patients with treatment-resistant depression: a candidate gene analysis. J Clin Psychiatry. 2012 Jun;73(6):878-85. doi: 10.4088/JCP.10m06744. Epub 2012 Mar 6. PMID 22480387
- [Derived] Houston J, Dharia S, Bishop JR, Ellingrod VL, Fijal B, Jacobson JG, Hoffmann VP. Association of DRD2 and ANKK1 polymorphisms with prolactin increase in olanzapine-treated women. Psychiatry Res. 2011 May 15;187(1-2):74-9. doi: 10.1016/j.psychres.2010.10.020. Epub 2010 Nov 20. PMID 21095016
- [Derived] Tohen M, Case M, Trivedi MH, Thase ME, Burke SJ, Durell TM. Olanzapine/fluoxetine combination in patients with treatment-resistant depression: rapid onset of therapeutic response and its predictive value for subsequent overall response in a pooled analysis of 5 studies. J Clin Psychiatry. 2010 Apr;71(4):451-62. doi: 10.4088/JCP.08m04984gre. Epub 2010 Feb 23. PMID 20361905
- [Derived] Thase ME, Corya SA, Osuntokun O, Case M, Henley DB, Sanger TM, Watson SB, Dube S. A randomized, double-blind comparison of olanzapine/fluoxetine combination, olanzapine, and fluoxetine in treatment-resistant major depressive disorder. J Clin Psychiatry. 2007 Feb;68(2):224-36. doi: 10.4088/jcp.v68n0207. PMID 17335320